CLINICAL TRIAL: NCT01540383
Title: From Controlled Experimental Trial to Everyday Communication: How Effective is Intensive Aphasia Therapy Under Routine Clinical Conditions?
Brief Title: Effectiveness of Intensive Aphasia Therapy Under Routine Clinical Conditions
Acronym: FCET2EC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Fresenius University of Applied Science (Other); Charite University, Berlin, Germany (Other); Entwicklungsgruppe Klinische Neuropsychologie, Klinikum Bogenhausen, München (Unknown); Institut für Biometrie und Klinische Epidemiologie, Charité Campus Benjamin Franklin, Berlin (Unknown); RWTH Aachen University (Other); Bundesverband für die Rehabilitation der Aphasiker e.V. (Unknown); Universitätsklinikum Leipzig (Other); MEDIAN Klinik Grünheide (Unknown); Brandenburgklinik Berlin-Brandenburg GmbH (Unknown); St. Mauritius Therapieklinik (Unknown); Aphasie- und Seniorenzentrum Josef Bergmann Vechta (Unknown); Behandlungs- und Rehabilitationszentrum für Intensiv-Therapie Lindlar (Unknown); Wickerklinik Bad Homburg v.d.H. (Unknown); Asklepios Neurological Clinic Falkenstein (Other); Akademische Praxis für Sprachtherapie / Praxis für Rehabilitationswesen Aschaffenburg (Unknown); Städtisches Klinikum München, Klinikum Bogenhausen (Unknown); Schoen Clinic Bad Aibling (Other); m&i-Fachklinik Bad Liebenstein (Unknown); m&i-Fachklinik Enzensberg (Unknown); m&i-Fachklinik Herzogenaurach (Unknown); mediclin Klinikum Soltau (Unknown); Moritz Klinik, Bad Klosterlausnitz (Unknown); Klinikum Christophsbad, Göppingen (Unknown); P.A.N.-Zentrum (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA1/234/11
Record Dates: First submitted 2012-02-06; First posted 2012-02-28 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Aphasia; Stroke
Keywords: Communication; Language; Treatment; Intervention; Therapy; Efficacy; Maintenance; Recovery; Outcome; Rehabilitation; Treatment Intensity; Language Impairment; Intensive Language Therapy; Functional Communication; Functional Improvement; Evidence-Based Intervention; High-Frequency
MeSH Terms: conditions — Aphasia; Stroke; Communication; Language; Language Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive aphasia therapy group (Experimental): Group starts intensive integrative aphasia therapy within 3 workdays (or as soon as possible) after baseline exam
  Interventions: Behavioral: Intensive integrative aphasia therapy
- Waiting list control group (Other): Group starts intensive integrative aphasia therapy after a waiting period of at least three weeks
  Interventions: Behavioral: Waiting list control group

INTERVENTIONS:
Behavioral: Intensive integrative aphasia therapy — Intensive language therapy (3 weeks, 5 days/week, >=2 hours/day) provided in regular clinical setting and consisting of a combination of language systematic and communicative-pragmatic treatment
  Arms: Intensive aphasia therapy group
Behavioral: Waiting list control group — Control group starts intensive language therapy after a 3-week waiting period.
  Arms: Waiting list control group

SUMMARY:
The purpose of this study is to examine whether 3 weeks of intensive language therapy provided in clinical in- and outpatient settings is effective in improving everyday communication in postacute/chronic post-stroke aphasia, as measured by performance on the Amsterdam Nijmegen Everyday Language Test (ANELT).

DETAILED DESCRIPTION:
Aims of the study:

This multicenter randomized placebo-controlled study aims to examine whether integrative intensive (> 10 hours/week for at least 3 weeks) language and communication therapy administered under routine clinical conditions translates into a statistically significant functional improvement of everyday communication in patients with chronic aphasia (i.e., aphasia persisting for 6 or more months after the stroke). A further aim is to examine whether therapy-induced improvements are still maintained over a period of six months. The study's results may lead to more targeted treatment regimens and thus to an enhancement of health-related quality of life in persons with chronic aphasia. The data will further provide evidence-based guidelines of best practice in the rehabilitation of persons with chronic aphasia.

Methods:

Fourteen in- and outpatient rehabilitation centres across Germany participate in the study. Via a digital randomization procedure, patients are allocated to one of two groups: an experimental group, starting as soon as feasible with treatment lasting 3 to 6 weeks, and a waiting list control group, whose therapy begins after a three-week delay. Both groups receive a combination of language systematic and communicative-pragmatic language therapy. Everyday language ability will be examined with a standardized outcome measure, and compared between groups at several points: immediately before as well as immediately after and 6 months after completion of (3-6 weeks) intensive language therapy.

Statistical analyses:

The primary analysis compares the changes in functional communication ability (as indicated by changes of pre- to post-therapy functional communication scores on the primary outcome measure, the ANELT) between the experimental and the waiting list control group in an intention-to-treat (ITT) design. To balance for unequal treatment durations across patient ("naturalistic treatment setting"), the critical pre- to post therapy interval is fixed at three weeks, with the option of extension of therapy (provided it is granted by the sickness fund) and re-test after termination of therapy. The long-term stability of potential treatment gains will be re-evaluated 6 months post therapy.

Further exploratory analyses will examine therapy-induced changes in secondary outcome measures (see below) in the experimental compared to the waiting list control group.

Considering that age, gender, time post stroke onset, aphasia type (fluent, non-fluent), aphasia severity (based on the Aachen Aphasia Test [AAT] profile score), the total hours of therapy provided, type of stroke (cortical strokes with or without subcortical involvement), the amount of therapy-concomitant self-administered language practice (e.g. computer-aided practice), and concurrent physio- and neuropsychological therapies might influence functional outcome, the above factors will be included in a multivariate analysis with variable selection. The amount of outpatient therapy provided after discharge from intensive treatment will be statistically controlled by covariate analyses.

Finally, the investigators expect that therapy effects in the waiting list control group will be comparable to those of the experimental group. Thus, after initiation of therapy in the control group after a three-week delay, outcome data will be collected in analogy to the experimental group, and will serve to replicate potential effects of intensive language therapy under routine clinical conditions.

ELIGIBILITY:
Inclusion Criteria:

* presence of aphasia for at least 6 months after non-hemorrhagic or hemorrhagic cortical or subcortical-cortical stroke
* native language German
* participant's comprehension ability needs to be sufficiently high to give informed consent
* participant's language abilities have to allow the administration of the Aachen Aphasia Test (AAT)

Exclusion Criteria:

* aphasia due to non-vascular etiology
* no evidence for aphasia (based on AAT subtests 'Token Test' and 'Written Language'
* severe untreated medical conditions which prohibit participation in intensive language therapy
* severe vision or hearing problems (uncorrected)
* participation in another interventional or language therapy study within four weeks before potential enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2012-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Changes on the Amsterdam Nijmegen Everyday Language Test (ANELT) - A-scale | Baseline is compared to performance immediately and 6 months post 3 weeks of intensive language therapy. Patients with at least 5 weeks of therapy, performance will also be assessed after therapy completion (on average 6 weeks)
  Mean gain in ANELT understandability scores (ANELT A-scale; using the parallel versions ANELT-I and ANELT-II)

SECONDARY OUTCOMES:
morbidity measure: changes in language-systematic aphasia screening (SAPS) | Baseline is compared to performance immediately and 6 months post 3 weeks of intensive language therapy. Patients with at least 5 weeks of therapy, performance will also be assessed after therapy completion (on average 6 weeks)
  Changes from pre- to post therapy of scores on:
  a (yet unpublished) test to assess language performance in 2 language modalities (perception, production) and 3 language levels (phonological, lexical, morphosyntactic). There are 3 different levels of complexity for each combination of modality and language level. Performance is thus assessed in 18 language domains (2x3x3).
morbidity measure: changes in communicative-pragmatic screening (KOPS) | Baseline is compared to performance immediately and 6 months post 3 weeks of intensive language therapy. Patients with at least 5 weeks of therapy, performance will also be assessed after therapy completion (on average 6 weeks)
  Changes from pre- to post therapy of scores on:
  an (yet unpublished) test measuring verbal and nonverbal performance in daily life communicative activities of increasing complexity
morbidity measure: changes in Modified Rankin Scale | Baseline is compared to performance immediately and 6 months post 3 weeks of intensive language therapy. Patients with at least 5 weeks of therapy, performance will also be assessed after therapy completion (on average 6 weeks)
  Changes from pre- to post therapy of scores in:
  the degree of disability or dependence in daily activities
quality of life measure: changes in German version of the Stroke and Aphasia Quality of Life Scale-39 (SAQOL-39) | Baseline is compared to performance immediately and 6 months post 3 weeks of intensive language therapy. Patients with at least 5 weeks of therapy, performance will also be assessed after therapy completion (on average 6 weeks)
  Changes from pre- to post therapy of scores on:
  Health-related quality of life questionnaire adapted for persons with aphasia
quality of life measure: changes in Communicative Effectiveness Index (CETI) and the ANELT partner communication questionnaire | Baseline is compared to performance 6 months post 3 weeks of intensive language therapy.
  Changes from pre- to post therapy of scores on:
  ratings of functional communication ability by relatives of persons with aphasia
morbidity measure: changes in nonverbal cognitive functions | Baseline is compared to performance immediately and 6 months post 3 weeks of intensive language therapy. Patients with at least 5 weeks of therapy, performance will also be assessed after therapy completion (on average 6 weeks)
  Changes from pre- to post therapy of scores on:
  * Nonverbal Learning Test (NVLT)
  * Trail Making Test
  * Verbal Fluency Test
quality of life measure: changes in Visual analog mood scales (VAMS) | Baseline is compared to performance immediately and 6 months post 3 weeks of intensive language therapy. Patients with at least 5 weeks of therapy, performance will also be assessed after therapy completion (on average 6 weeks)
  Changes from pre- to post therapy of scores on:
  assessment of mood visual analog scales (adapted for persons with aphasia)
changes in Amsterdam-Nijmegen Everyday Language Test (ANELT) - B-scale | Baseline is compared to performance immediately and 6 months post 3 weeks of intensive language therapy. Patients with at least 5 weeks of therapy, performance will also be assessed after therapy completion (on average 6 weeks)
  Mean gain in ANELT intelligibility scores (ANELT B-scale; using the parallel versions ANELT-I and ANELT-II)
changes in Amsterdam-Nijmegen Everyday Language Test (ANELT) - syntactic rating | Baseline is compared to performance immediately and 6 months post 3 weeks of intensive language therapy. Patients with at least 5 weeks of therapy, performance will also be assessed after therapy completion (on average 6 weeks)
  Mean gain in syntactic rating scores (syntax rating criteria based on AAT subtest "spontaneous speech") for the ANELT scenarios (using the parallel versions ANELT-I and ANELT-II)
changes in Amsterdam-Nijmegen Everyday Language Test (ANELT) - nonverbal communication rating | Baseline is compared to performance immediately and 6 months post 3 weeks of intensive language therapy. Patients with at least 5 weeks of therapy, performance will also be assessed after therapy completion (on average 6 weeks)
  Mean gain in nonverbal rating scores (criteria based on "Scenario Test") for the ANELT scenarios (using the parallel versions ANELT-I and ANELT-II)

CONTACTS AND LOCATIONS:
Overall Officials: Annette Baumgaertner, PhD, Principal Investigator — Hochschule Fresenius University of Applied Science; Caterina Breitenstein, PhD, Principal Investigator — Neurology, University of Muenster; Agnes Floel, MD, Study Director — Neurology, Universitätsmedizin Charite, CCM, Berlin; Wolfram Ziegler, PhD, Principal Investigator — Clinical Neuropsychology Research Group (EKN), Klinikum Bogenhausen, München; Tanja Grewe, PhD, Principal Investigator — Hochschule Fresenius University of Applied Sciences
Locations (1):
- University of Muenster, Münster, North Rhine-Westfalia, Germany

REFERENCES:
- [Derived] Breitenstein C, Grewe T, Floel A, Ziegler W, Springer L, Martus P, Huber W, Willmes K, Ringelstein EB, Haeusler KG, Abel S, Glindemann R, Domahs F, Regenbrecht F, Schlenck KJ, Thomas M, Obrig H, de Langen E, Rocker R, Wigbers F, Ruhmkorf C, Hempen I, List J, Baumgaertner A; FCET2EC study group. Intensive speech and language therapy in patients with chronic aphasia after stroke: a randomised, open-label, blinded-endpoint, controlled trial in a health-care setting. Lancet. 2017 Apr 15;389(10078):1528-1538. doi: 10.1016/S0140-6736(17)30067-3. Epub 2017 Mar 1. PMID 28256356
- [Derived] Baumgaertner A, Grewe T, Ziegler W, Floel A, Springer L, Martus P, Breitenstein C. FCET2EC (From controlled experimental trial to = 2 everyday communication): How effective is intensive integrative therapy for stroke-induced chronic aphasia under routine clinical conditions? A study protocol for a randomized controlled trial. Trials. 2013 Sep 23;14:308. doi: 10.1186/1745-6215-14-308. PMID 24059983